CLINICAL TRIAL: NCT07165912
Title: Effects of a Group Versus Individual Cognitive Training Program on Chemotherapy-induced Cognitive Impairment (Chemobrain) in Breast Cancer Patients Undergoing Active Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Juan Luis Sanchez Gonzalez, Dr., University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ChemoSala
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Females; Oncology
Keywords: Cognitive training; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group intervention (Experimental): The program is organized into four progressive months: (1) cognitive and emotional security, with activities focused on attention, basic memory, and group bonding; (2) flexibility and problem solving, where executive functions, language, and personal narrative are stimulated; (3) cognitive challenges and emotional control, which strengthen spatial memory, self-concept, and relaxation techniques; and (4) closure and consolidation of learning, dedicated to reinforcing achievements, promoting gratitude, and strengthening mutual support. In this way, ALMA not only seeks to train the mind, but also to provide a space for comprehensive support for the emotional and physical well-being of the participants.
  Interventions: Behavioral: Health Education Program
- Individual intervention group (Experimental): The indiviudal cognitive training program (CT) focused on everyday cognition (EC) will be conducted individually. Each participant will receive a dossier specifically designed for the study.
  The intervention will consist of four training periods over a duration of 4 months (Period 1, P1; Period 2, P2; Period 3, P3; Period 4, P4), with 20 activities each. Each period will last one month (5 activities per week).
  Interventions: Behavioral: Group training program
- Health Education Program (Active Comparator): Instructions and recommendations will be provided in an informative leaflet to promote an active and healthy lifestyle, encouraging self-care and good practices. This leaflet will include the new WHO guidelines, which recommend specific measures to reduce the risk of cognitive decline. These measures are: Eating healthy foods, engaging in physical activity, maintaining social connections, playing challenging cognitive games, getting good sleep, managing stress, staying hydrated, and avoiding smoking and excessive alcohol consumption.
  Interventions: Behavioral: Individual Cognitive Training Program

INTERVENTIONS:
Behavioral: Health Education Program — An informative leaflet will promote a healthy lifestyle with WHO guidelines to reduce cognitive decline, recommending a balanced diet, physical activity, social engagement, cognitive games, good sleep, stress management, hydration, and avoiding smoking and excessive alcohol.
  Arms: Group intervention
Behavioral: Individual Cognitive Training Program — The cognitive training program (CT) on everyday cognition (EC) will be individualized, with each participant receiving a tailored dossier. The intervention includes four 1-month training periods (P1-P4), each featuring 20 activities, conducted at a rate of 5 activities per week over 4 months.
  Arms: Health Education Program
Behavioral: Group training program — The group cognitive training program (CT) on everyday cognition (EC) will be individualized, with each participant receiving a tailored dossier. The intervention includes four 1-month training periods (P1-P4), each featuring 20 activities, conducted at a rate of 5 activities per week over 4 months.
  Arms: Individual intervention group

SUMMARY:
Introduction: The significant improvement in breast cancer survival, largely attributable to biomedical and technological progress, makes it increasingly necessary to investigate the secondary effects linked to this pathology. Among these, cancer-related cognitive impairment (CRCI) stands out as one of the most frequent yet frequently overlooked complications.

Objective: To evaluate the impact of a structured cognitive training program on the management of CRCI in patients with breast cancer receiving active treatment.

Methodology: A randomized controlled clinical trial will be conducted with two arms: an Intervention Group (IG) and a Control Group (CG). The study will include patients with a recent diagnosis of breast cancer. Based on sample size calculations, 50 participants will be recruited-25 per group-to detect a minimum difference of 2.95 points on the MoCA (Montreal Cognitive Assessment), a tool commonly used to assess cognitive performance. All participants will receive an informational leaflet aligned with the latest WHO recommendations for preventing cognitive decline. In addition, the IG will complete an individualized cognitive training (CT) program focused on everyday cognitive skills (EC). The program will provide a dossier with 80 training sessions, structured into four phases (P1-P4) of 20 activities each, to be implemented monthly. Baseline assessments and a follow-up four months after the intervention will be carried out in both groups. Variables collected will include sociodemographic and clinical data, as well as outcome measures for cognitive status (MoCA), everyday cognition (PECC), anxiety levels (Hamilton scale), functional capacity (LB), sleep quality (PSQI), quality of life (ECOG), and subjective memory complaints (FACT-COG).

Impact: Findings from this study could support the development of targeted cognitive rehabilitation strategies and the implementation of clinical protocols for individuals undergoing breast cancer treatment. By addressing CRCI-an underrecognized but increasingly prevalent issue given rising survival rates-these interventions may contribute to improving patients' overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

Being an adult (18 years or older). Having a recent histopathological diagnosis of newly diagnosed breast cancer and starting oncological treatment.

Being fully capable of performing daily functions. Willingness to voluntarily participate in the study and signing the informed consent.

Exclusion Criteria:

Lack of literacy skills or significant language comprehension deficit. Diagnosis of a Central Nervous System tumor or participation in another cognitive stimulation program.

Clinical diagnosis of a neurocognitive disorder as defined in the DSM-V.

Withdrawal Criteria:

Dropping out of the program or not completing the final evaluation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | Baseline; "4 months final"
  The Montreal Cognitive Assessment Test (MoCA Test) Version 8.3. This test detects mild cognitive impairment (MCI) by assessing executive functions, attention, abstraction, memory, calculation, and orientation. It takes about 10 minutes to administer. The maximum score is 30 points, with scores below 26 indicating MCI
Subjective Perception of Cognitive Impairment in Cancer Patients | Baseline; "4 months final"
  FACT-COG (Version 3) (24): This 37-item questionnaire is divided into six cognitive domains: memory, concentration, mental acuity, verbal fluency, functional interference, and multitasking ability. Additionally, it includes two subscales: "notability" (comments from others) and "perceived impact of cognitive impairment on quality of life." Respondents indicate the frequency of each occurrence over the past 7 days on a 5-point Likert scale, from 0 ("never") to 4 ("several times a day"). The scores from the individual subscales are summed to determine the total FACT-Cog score, ranging from 0 to 148, with higher scores indicating better cognitive functioning.

SECONDARY OUTCOMES:
Everyday Cognition | Baseline; "4 months final"
  Test for the Evaluation of Everyday Cognition (PECC) (18): This test measures an individual's ability to solve 12 real-life situations in areas such as medication management, administrative tasks, financial management, meal preparation, transportation, and shopping, thus assessing functional capacity in daily life. The administration time is 35 minutes.
Anxiety | Baseline; "4 months final"
  Hamilton Anxiety Rating Scale (19): A clinical assessment tool used to measure the level of anxiety experienced by a person. It consists of 14 items, each with five response options ranging from "not present" to "very severe." The final score can be 17 or less (mild anxiety), between 18 and 24 (moderate anxiety), and between 25 and 30 (severe anxiety).
Functionality | Baseline; "4 months final"
  Lawton and Brody Instrumental Activities of Daily Living (IADL) Scale (20): Designed to evaluate autonomy in instrumental activities in older adults. It takes about 4 minutes to administer, scoring each item as 0 or 1, with a total score of 8.
Sleep Quality | Baseline; "4 months final"
  Pittsburgh Sleep Quality Index (PSQI) (21): Designed to measure sleep quality in individuals aged 24 to 83 years. It takes 5-10 minutes to administer. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Subjective Memory Failures | Baseline; "4 months final"
  Everyday Memory Failures Questionnaire (23): It includes categories such as "talking, reading, and writing," "names and faces," "actions," and "learning new things." Responses are given on a 9-point Likert scale, ranging from "Not at all in the last 3 months" to "More than once a day." Due to the complexity of the nine options, some authors use fewer response options.

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Luis, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon request in the GREDOS scientific repository of the University of Salamanca once the study is completed. Link: https://gredos.usal.es/handle/10366/3823.
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: The data will be available upon request in the GREDOS scientific repository of the University of Salamanca once the study is completed. Link: https://gredos.usal.es/handle/10366/3823.